CLINICAL TRIAL: NCT00574964
Title: Phase II Treatment of Adults With Newly Diagnosed Supratentorial Glioblastoma Multiforme Treated With Gliadel Wafers, Surgery and Limited Field Radiation Plus Concomitant Temozolomide Followed by Temozolomide
Brief Title: Gliadel Wafers and Temodar in the Treatment of Glioblastoma Multiforme
Acronym: Temodar
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institution.
Sponsor: University of Iowa (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Timothy Ryken, MD, University of Iowa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200408035
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2010-03

CONDITIONS: Primary Glioblastoma Multiforme
MeSH Terms: interventions — Carmustine; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Gliadel Wafer, Temodar and Radiotherapy

INTERVENTIONS:
Other: Gliadel Wafer, Temodar and Radiotherapy — Given concurrently starting 10-30 days after surgery.

SUMMARY:
The purpose of this research study is to determine if combining all three treatments of Gliadel wafers, Temozolomide and Radiation therapy at the same time is safe and more effective than one treatment at a time. The study will measure the survival of subjects treated with this combination of drugs.

DETAILED DESCRIPTION:
Subjects will receive surgery + Gliadel® wafer implantation + Limited Field Radiation Therapy to a dose of 61.2 Gy with concomitant daily temozolomide. Up to 8 wafers will be implanted into the tumor resection cavity (depending upon its size) after maximal tumor resection. Between days 10 and 30 all subjects will begin a standard course of post-operative limited field radiation therapy to the tumor site and a surrounding margin, with concomitant daily temozolomide (75mg/m2 x 7 d/wk for 6 weeks, concomitant chemoradiotherapy phase). Beginning no later than 45 days following completion of radiation, temozolomide will be given at a dosage of 200 mg/m2 daily for five days on a 28 day schedule, for a total of 6 cycles (adjuvant chemotherapy phase). Subjects will be monitored weekly during chemoradiotherapy with CBC with differential and brief clinical assessment, and monthly during the adjuvant chemotherapy phase. Toxicity reports will be assessed every three months. Dose limiting toxicities (DLT) are defined in section 4.2. If toxic events unresponsive to planned dose modification exceed 20% of enrolled subjects the stopping rule will be met and the study will be discontinued. MRIs will be obtained no more than 72 hours post-op, and then prior to the first, third, and fifth cycles of monthly temozolomide. Additionally, a stealth MRI or CT scan (with or without contrast) will be done one week prior to radiotherapy for treatment planning at the discretion of the treating Radiation Oncologist. Following completion of the entire course of treatment subjects will be monitored clinically as well as with MRI every 3 months for survival and evidence of progression.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Subjects must have findings on neuroimaging studies and clinical evaluation consistent with the diagnosis of a primary brain tumor in order to be offered enrollment in the study. Subsequently, in order to remain on study, they must have histologically or cytologically confirmed primary tumor of the brain. Intra-operative confirmation of histology (i.e. frozen section assessment or equivalent) is required for all subjects. Gliadel wafers will not be implanted without positive intraoperative histopathology consistent with a primary tumor of the brain. The final classification and evaluability determination will be made based on post-operative histological reports showing anaplastic astrocytoma or Glioblastoma multiforme. No central pathology review will be required.
* Newly diagnosed supratentorial primary brain lesion as visualized on enhanced MRI scan (or CT scan with contrast for subjects who cannot undergo MRI) that is appropriate for surgical resection and implantation of Gliadel.
* All eligible subjects will undergo surgical resection. After resection, if there is communication of the resection cavity with the ventricular spaces preventing the use of Gliadel® the subject leaves the study.
* MRI or CT with and without contrast within 30 days of study entry.
* New diagnosis of primary brain tumor is required. No prior therapy, including previous radiotherapy, chemotherapy, or operation is allowed.
* Age 18 years and older, since the rationale for this therapy was established in adults, and the tumor uncommon in children, so that no useful information is likely to emerge from their inclusion in this study.
* Karnofsky Performance Status greater than or equal to 60.
* Life expectancy of at least 12 weeks.
* Subjects must have normal organ and marrow function as defined below:

  * WBC greater than or equal 2,000/mm3
  * Absolute neutrophil count greater than or equal to 1,500/mm3
  * Platelets greater than or equal to 125,000/mm3
  * Total bilirubin less than or equal to 2.0 mg/dl
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X upper limit of normal
  * PT / PTT within 1.5 X upper limit of normal
  * Creatinine less than or equal to 1.7 mg/dl
  * BUN less than or equal to 40 mg/dl
  * Hemoglobin > 10 g/dL
* Clinical evaluation of cardiac and pulmonary functions consistent with adequate tolerance of surgical procedure.
* Negative pregnancy test (beta HCG) if a female of childbearing age and not surgically sterilized.
* The effects of BCNU (the active ingredient in the Gliadel wafer) with concomitant Temozolomide on the developing human fetus are unknown. BCNU is known to cause fetal harm if administered to a pregnant woman and is a pregnancy risk factor D. Temozolomide May cause fetal harm when administered to pregnant women. Animal studies, at doses less than used in humans, resulted in numerous birth defects. Testicular toxicity was demonstrated in animal studies using smaller doses than recommended for cancer treatment. Temozolomide is also a pregnancy risk factor D. Radiation therapy is known to be both mutagenic and teratogenic. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, or if her partner is participating in this trial, she should inform the treating physician immediately.

Exclusion Criteria:

* Known hypersensitivity or allergy to BCNU (carmustine) or other components of the Gliadel® wafer such as polifeprosan polymer.
* Known hypersensitivity to temozolomide.
* Subjects may not be receiving any other investigational agents.
* If the surgeon determines that placement of Gliadel wafers is inappropriate, or if the final diagnosis is other than anaplastic astrocytoma or glioblastoma, the subject will leave the study and not be further analyzed.
* Subjects who have had chemotherapy or radiotherapy at any time for this diagnosis.
* A subject will be considered unresectable preoperatively if, in the opinion of the neurosurgeon, the subject is not a candidate for maximal cytoreductive surgery, (i.e., crosses the midline, continuous with the ventricular space). Such subjects will not be eligible for treatment on this protocol.
* Diagnosis of prior central nervous system tumor.
* Diagnosis of systemic cancer requiring treatment within the past five years (except for non-melanotic carcinoma of the skin or carcinoma in situ of the cervix).
* Open communication of the resection cavity with the ventricular system that prevents insertion of Gliadel or tumors that cross the midline.
* Posterior fossa or brain stem tumor.
* Concurrent severe medical illness (e.g., active infection, acute hepatitis, cardiac arrhythmia, unstable angina, congestive heart failure, uncontrolled diabetes mellitus, uncontrolled seizures, pulmonary insufficiency, pulmonary fibrosis, pulmonary embolus, etc) or psychiatric illness, or abnormal laboratory values that preclude surgical candidacy or limits expected survival to less than 12 weeks.
* Pregnant women are excluded from this study because BCNU and/or Temozolomide are pregnancy risk D pharmaceutical agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BCNU and/or Temozolomide, breastfeeding should be discontinued if the mother is treated with either of these agents. These potential risks may also apply to other agents used in this study.
* Subjects with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive subjects receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with BCNU or other agents administered during the study. Appropriate studies will be undertaken in subjects receiving combination anti-retroviral therapy when indicated.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety and feasibility of Gliadel 3.85% wafers plus surgery and limited field radiation therapy with concomitant temozolomide, followed by adjuvant temozolomide, in subjects undergoing initial surgery for newly-diagnosed malignant gliomas. | Will follow subjects to collect DOD.

SECONDARY OUTCOMES:
Determine the progression free survival at 6 months, medial survival, and one year survival rate of this subject population. Determine objective response rate. | Will follow subject to collect DOD.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Ryken, MD, Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Clinic, Iowa City, Iowa, United States